CLINICAL TRIAL: NCT02100111
Title: RONNIE - A Multi-Center, Multi-National, Retrospective Medical Record Review to Describe Treatment Patterns and Outcomes for Patients With Locally Advanced or Metastatic Basal Cell Carcinoma
Brief Title: An Analysis of Treatment Patterns and Outcomes for Basal Cell Carcinoma (BCC) Cancer Participants
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: MO28682
Record Dates: First submitted 2014-03-20; First posted 2014-03-31 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-06

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with advanced or metastatic BCC: Participants with BCC who received any treatment including surgeries, radiation, photodynamic therapy, chemotherapy, supportive/palliative care, or other therapies, will be included as a part of study.

SUMMARY:
This multi-center, observational study involves reviewing the medical records of approximately 100 adult participants diagnosed with advanced BCC from 01 January 2005 until 31 December 2010. Participant records will be analyzed to identify participant characteristics, treatment patterns and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of advanced BCC, defined as (1) locally advanced BCC (inoperable as determined by the site investigator or surgery contraindicated) with receipt of radiation therapy (unless radiation was contraindicated), or (2) metastatic BCC, from 01 January 2005 through 31 December 2010

Exclusion Criteria:

* Participation in an interventional trial that dictated treatment during the study time period (01 January 2005 - 31 December 2010), or within 90 days prior to individual participant' study enrolment dates
* Participants undergoing treatment with a Hedgehog pathway inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with locally advanced or metastatic BCC
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2011-12-31 (Actual)

PRIMARY OUTCOMES:
Participants Demographics: Age at Initation of Study | Baseline (Initiation of the study)
Participants Demographics: Gender at Initation of Study | Baseline
Participants Demographics: Race at Initation of Study | Baseline
Participants Demographics: Country of Enrollment at Initation of Study | Baseline
Percentage of Participants Categorized as per BCC Disease History | Baseline up to 9 months
Percentage of Participants Categorized as per BCC Type | Baseline up to 9 months
Percentage of Participants Categorized as per Site of Primary Lesion | Baseline up to 9 months
Percentage of Participants Categorized as per Number of Lesions | Baseline up to 9 months
Percentage of Participants Categorized as per Size of Lesions | Baseline up to 9 months
Percentage of Participants Categorized as per Histopathology of BCC | Baseline up to 9 months
Percentage of Participants Categorized as per Basal Cell Carcinoma Nevus Syndrome (BCCNS) Status | Baseline up to 9 months
Percentage of Participants Categorized as per Eastern Cooperative Oncology Group (ECOG) Performance Status | Baseline up to 9 months
Percentage of Participants Categorized as per Number of Biopsies Undergone | Baseline up to 9 months
Percentage of Participants Categorized as per Type of BCC Treatment Received | Baseline up to 9 months
Percentage of Participants With Complete Response | Baseline up to 9 months
Percentage of Participants With Partial Response | Baseline up to 9 months
Percentage of Participants With Stable Disease | Baseline up to 9 months
Percentage of Participants With Disease Progression | Baseline up to 9 months
Percentage of Participants Who Died | Baseline up to event of death assessed maximum up to 9 months
Percentage of Participants With Progression Free survival | Baseline up to 9 months
Percentage of Participants Categorized as per Impact of Surgery for BCC on Organ Function | Baseline up to 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (42):
- France (25):
  - Hotel Dieu; Dermatologie, Angers
  - Hopital Prive D Antony; Dermatologie, Antony
  - Hôpital St Jacques de Besançon; (Dermatology), Besançon
  - Hopital Saint Andre CHU De Bordeaux; Dermatologie, Bordeaux
  - Hopital Ambroise Pare; Sce Dermatologie, Boulogne-Billancourt
  - Hopital La Cavale Blanche; Medecine 1, Brest
  - Chu Estaing; Dermatologie, Clermont-Ferrand
  - Hopital Victor Jousselin; Dermatologie, Dreux
  - Chi Emile Durkheim Site Epinal; Oncologie, Épinal
  - Hôpital Albert Michallon; Derm Phlebologie Allergologie, Grenoble
  - Hopital Saint Vincent; Consult Dermatologie Enfants, Lille
  - Hopital Claude Huriez; Sce Dermatologie, Lille
  - Hopital Dupuytren; Dermatologie, Limoges
  - Hopital Timone Adultes; Radiotherapie Oncologie, Marseille
  - Hopital Jacques Monod; Dermatologie, Montivilliers
  - Hopital Saint Eloi; CHU de Montpellier; Svc de Dermatologie, Montpellier
  - Hopital Bichat Claude Bernard; Sce Dermatologie, Paris
  - Hopital Saint Louis; Dermatologie 1, Paris
  - Hopital de Haut-Leveque; Dermatologie Serv., Pessac
  - Centre Hospitalier Lyon Sud; Dermatologie, Pierre-Bénite
  - Chu La Miletrie; Dermatologie, Poitiers
  - Hopital Laennec; Sce Dermatologie, Quimper
  - Hopital Nord ; Dermatologie, Saint-Etienne
  - Hopital Sud; Dermatologie, Salouël
  - Hopitaux de Brabois; Dermatologie, Vandœuvre-lès-Nancy
- Germany (8):
  - HELIOS Klinikum Erfurt, Klinik für Hautkrankheiten und Allergologie, Erfurt
  - Klinik Johann Wolfgang von Goethe Uni; Klinik für Dermatologie, Venerologie und Allergologie, Frankfurt
  - SRH Wald-Klinikum Gera; Klinik für Hautkrankheiten und Allergologie, Gera
  - Universitätsmedizin Greifswald; Klinik für Mund-Kiefer-Gesichtschirurgie/Plastische Operationen, Greifswald
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz KöR, Hautklinik und Poliklinik, Mainz
  - Klinikum Mannheim Klinik fuer Dermatologie, Venerologie und Allergologie, Mannheim
  - Klinikum der LMU München; Klinik und Poliklinik für Dermatologie und Allergologie, München
  - Klinikum Dorothea Ch.Erxleben; Klinik für Dermatologie und Allergologie, Quedlinburg
- Italy (7):
  - Irccs Crob, Rionero in Vulture, Basilicate
  - Arcispedale Santa Maria Nuova; Dermatologia, Reggio Emilia, Emilia-Romagna
  - Spedali Civili di Brescia, Brescia, Lombardy
  - Università del Piemonte Orientale; Dipartimento di Dermatologia, Novara, Piedmont
  - Policlinico Le Molinette; Clinica Dermatologica, Turin, Piedmont
  - Azienda Sanitaria di Firenze Presidio Palagi - SC Dermatologia II e Fisioterapia Dermatologica, Florence, Tuscany
  - A.O. Univ. Senese Policlinico S. Maria alle Scotte; Dip. Medicina clinica e Scienze Immunologiche, Siena, Tuscany
- United Kingdom (2):
  - Western Infirmary; Division of Cardiovascular and Medical Sciences, Glasgow
  - Manchester Royal Infirmary; Department Of Medicine, Manchester